Title: Comparing right colon adenoma and hyperplastic polyp miss rate in

colonoscopy using water exchange and carbon dioxide insufflation: A prospective

randomized controlled trial

INTRODUCTION

Colonoscopy is currently regarded as the gold standard to detect and prevent

colorectal cancer (CRC) [1]. It estimated to prevent about 76%-90% of CRC [2], but

post-colonoscopy CRCs (PCCRCs) still occur. Recent case-control studies consistently

demonstrated that protection by colonoscopy against right-sided colon cancer,

ranging from 40% to 60%, was lower than the 80% protection attained in the left

colon [3-5]. Of all PCCRCs, 58% were attributed to lesions missed during examination

[6]. In a systematic review of tandem colonoscopy studies, a 22% pooled miss-rate

for all polyps was reported [7]. Colonoscopy maneuvers helping to reduce miss-rate

for all polyps, particularly in the right colon, have the potential to decrease the

incidence of PCCRCs.

Water exchange (WE) colonoscopy is characterized by the gasless insertion to the

cecum in clear water and maximizing cleanliness during insertion. WE colonoscopy

has been shown to improve the overall adenoma detection rate (ADR), compared to

air insufflation colonoscopy, in many prospective randomized controlled trials (RCTs)

[8-13]. WE colonoscopy also has been shown to improve right colon ADR in RCTs

[10-12] and meta-analyses [14,15]. In a pooled data from two multisite RCTs, WE also

significantly increases right colon combined advanced and sessile serrated ADR as

compared to air insufflation colonoscopy [16]. Decreased multitasking-related

distraction from cleaning maneuvers has been the most recently identified

explanation for the increase in ADR by WE [17]. The right colon is usually the worst

prepared segment and proximal colorectal neoplasms with advanced histology

頁 1/13

frequently are smaller than the ones in the left colon or have a nonpolypoid

appearance [18,19]. Therefore, the adoption of WE in the right colon might be

especially beneficial.

Traditionally, all CRC are believed to arise from the adenomas through the

adenoma-carcinoma sequence. However, recent studies showed that 35% of CRC

were derived from serrated lesions (SLs) [20], which include hyperplastic polyp (HP),

sessile serrated adenomas/polyps (SSA/Ps) and traditional serrated adenomas [21].

The presence of SLs, even small and diminutive proximal HPs, has been reported to

be associated with higher rates of synchronous advanced neoplasia [22,23]. Proximal

HPs might also serve as precursors of cancer through DNA methylation and deficient

DNA mismatch repair [24-26]. However, SLs tend to be pale and flat and pose a

challenge for the endoscopists to detect them [27]. WE might come in handy for

uncovering the proximal SLs through the above stated mechanisms.

The primary outcome of this study is the right colon combined adenoma miss rate

(AMR) and hyperplastic polyp miss rate (HPMR) determined by tandem inspection of

the right colon using WE or CO2 insufflation for screening, surveillance, or positive

fecal immunochemical test (FIT) indications. The secondary outcomes are the overall

ADR and other adenoma detection related metrics between the two colonoscopy

methods.

**METHODS** 

This will be a prospective RCT comparing CO2 insufflation and WE in terms of right

colon combined AMR and HPMR by tandem inspection. It is originally designed as a

multicenter study conducted in three community hospitals in Taiwan. Consecutive

patients will be enrolled from April 2019 to October 2020. A written informed

consent will be obtained from all participating patients. The study has obtained

頁 2/13

ethical approval from the Joint Institutional Review Board of Taiwan (19-002-T-1) and

has been registered with ClinicalTrials.qov (NCT03845933). Due to delay in obtaining

IRB approval in two of the participating hospitals (Dalin Tzu-Chi Hospital obtained IRB

approval in late May 2019 and has not recruited any patient; Taipei Medical

University Hospital has not obtained IRB approval in early June 2019) and rapid

recruitment of Evergreen General Hospital since April 2019, which has recruited and

completed more than 90 patients in the end of May 2019, we have amended the

study design from multicenter study to single center study and have obtained the

approval of this amendment on July 19, 2019 from the Joint Institutional Review

Board of Taiwan.

**Participants** 

Consecutive patients aged 45 years or older undergoing colonoscopy for screening,

surveillance, and positive FIT will be considered for enrollment [28]. Exclusion criteria

will include familial adenomatous polyposis and hereditary non-polyposis CRC

syndrome, personal history of CRC or inflammatory bowel disease, previous colonic

resection, obstructive lesions of the colon, gastrointestinal bleeding, allergy to

fentanyl or midazolam, American Society of Anesthesiology (ASA) classification of

physical status grade 3 or higher (e.g. controlled congestive heart failure, stable

angina, previous heart attack, poorly controlled hypertension, morbid obesity,

chronic renal failure, bronchospastic diseases with intermittent symptoms), mental

retardation, pregnancy, and refusal to provide a written informed consent.

Randomization

Patients will be randomized in a 1:1 ratio to undergo either the CO2 insufflation

colonoscopy (CO2 group) or WE colonoscopy (WE group). Randomization will be

carried out by a computer-generated random sequence. Stratification based on

頁 3/13

colonoscopists and colonoscopy indications (screening, surveillance, and positive FIT)

will be performed. Individual random sequence will be placed in an opaque envelope

kept by an independent research assistant not directly involved in this study, which

will be opened immediately before the procedure.

**Bowel Preparation and Sedation** 

Patients will be instructed to eat low-residual foods for two days before

colonoscopy. Oral and written instructions on the split-dose bowel preparation

(Polyethylene glycol solution) will be provided to all patients. Colonoscopy will be

performed without sedation or with moderate sedation (intravenous fentanyl plus

midazolam). Moderate sedative agents will be administered by endoscopists.

**Colonoscopy Procedures** 

Colonoscopies will be performed by two board-certified colonoscopists (Chi-Liang

Cheng, Yen-Lin Kuo). Standard colonoscopes (CF-Q260AL/I; Olympus Medical Systems

Corp., Tokyo, Japan) will be used. All colonoscopists have performed more than 1000

conventional colonoscopies. Hands-on coaching by a WE expert (Felix W. Leung) to

standardize the WE method has been completed. Each colonoscopist has or will have

completed 100 cases of WE learning curve. Felix W. Leung will be involved in the

study design, data analyses, and report preparation, but not in patient enrollment. All

the colonoscopic procedures will be recorded.

Antispasmodic medication will not be administered during colonoscopy

examination. CO2 insufflation will be used for CO2 group and the withdrawal phase

of the WE group. Colonoscopy will begin with the patients in the left lateral position.

In the WE group, the air pump will be turned off before starting the procedure.

During the insertion phase, air and residual water or feces in the rectum will be

aspirated, and then the colon will be irrigated with warm water (32C-35C) using

flushing pumps (Olympus AFU-100; Olympus Corp.). There will be no restriction placed on the overall volume of water infused to achieve adequate cleansing. Suction and infusion of water will be performed sequentially because the endoscope has only one channel. Air pockets, when encountered, will be aspirated. When the cecum is reached and after most of the water is suctioned to collapse the cecal lumen, CO2 will be opened. In the CO2 group, colonoscopy is performed in the usual fashion, with minimal insufflation required to aid insertion. Cleaning in the CO2 group will be performed entirely during withdrawal. In the CO2 group, suction marks will be deliberately produced in the hepatic flexure and cecum to mimic the same marks frequently produced by the WE technique. Cecal intubation will be defined as the passage of the scope tip beyond the ileocecal valve with visualization of the medial wall between the ileocecal valve and the appendix orifice.

Upon arriving at the cecum, CO2 insufflation will be used in both groups and the scope will be withdrawn from the cecum to the hepatic flexure, with inspection of the mucosa at the same time. All polyps identified will be resected and sent for pathology evaluation. The most distal part of the hepatic flexure will be marked by a forceps biopsy and then the scope will be reinserted into the cecum by the first endoscopist using CO2 insufflation. A tandem inspection of the right colon will then be performed by a second endoscopist blinded to the insertion method in both study groups. All polyps found herein will be counted as the missed polyps. After the second withdrawal to the mark of distal hepatic flexure, the remainder of the colon will be examined in a standard manner by the first endoscopist. To assess the adequacy of blinding, the second endoscopist will be asked at the end of tandem right colon examination to guess which insertion method has been used. If less than 66% of these answers are correct, then adequate blinding will be considered to have

Date: 07/19/2019

been achieved.

Polyp search and resection will be performed during the withdrawal phase in both

groups. Insertion polypectomy will not be performed. All proximal colon polyps will

be removed irrespective of their size and appearance. All diminutive polyps with

hyperplastic appearance (based on narrow band imaging) in the rectosigmoid colon

will be documented by photography and left alone. Polyp size will be determined by

comparison with an opened biopsy forceps or a snare.

In both groups, the following information will be recorded: bowel preparation

quality using the Boston Bowel Preparation Scale (BBPS) score [29]; the total amount

of sedative medications (in procedures with sedation); the length of colonoscopy

reaching cecum; the amount of water infused and suctioned during insertion and

withdrawal phases; the procedure time taken for insertion and withdrawal for the

first examiner; the procedure time taken for tandem right colon inspection; the need

of abdominal compression and/or positon change to assist colonoscopy insertion;

the overall polyp number, size, histology and location; the missed right colon polyp

number, size, histology and location.

**Definition** 

Screening colonoscopy will be defined as either asymptomatic patients undergoing

their first colonoscopic examination or patients with a history of negative screening

colonoscopy undergoing their 5-year or 10-year follow-up examinations. Surveillance

colonoscopy will be defined as patients with a history of colon polyps undergoing

their follow-up examinations. Complete colonoscopy will be defined as successful

cecal intubation. Insertion time will be defined as the time between the scope

insertion and cecal intubation. Three stopwatches will be used to record the time

taken for mucosal cleaning (water infusion and suction), mucosal inspection, and

頁 6/13

polyp treatment respectively. Withdrawal time will be defined as the time from cecal intubation to the time when the colonoscope is withdrawn from the anus, including the time taken for mucosal cleaning, mucosal inspection, polyp biopsy and polypectomy. Total procedure time will be the sum of insertion time and withdrawal time. Three stopwatches will be used to record the time taken for mucosal cleaning, mucosal inspection, and polyp treatment, respectively, during the tandem right colon examination. Total duration of tandem right colon examination will be defined as the time of repeated examination from cecum to hepatic flexure by the blinded examiner, including the time taken for mucosal clearing, inspection and polyp treatment. Near-complete removal of infused water during insertion of WE is defined as ≥90% removal of infused water. Inspection times by the first and second endoscopists will be recorded. Comparable inspection times in the study and control groups will support the use of equivalent withdrawal inspection methods.

All colonic polyps removed during procedures will be sent for histological examination with clear labeling of location and sequences of colonoscopy. The location of colonic polyps will be defined according to the anatomical distribution. Right colon will be defined as cecum, ascending colon, and hepatic flexure. Proximal colon will be defined as right and transverse colon. Diminutive polyps will be defined as polyps with size ≤5 mm. Small polyps will be defined as polyps with size 6-9 mm. Large polyps will be defined as polyps with size ≥10 mm. Adenomas will include all adenomas and sessile serrated adenoma. Advanced adenomas will be defined as those lesions with one of the following criteria: 1) lesions larger than 10 mm in diameter; 2) lesions with a villous component; 3) lesions with high-grade dysplasia; and 4) lesions with invasive features.

ADR will be defined as the proportion of colonoscopies with at least one adenoma.

Advanced ADR will be defined as the proportion of colonoscopies with at least one

advanced adenoma. Mean adenoma per procedure (MAP) will be defined as the total

number of adenomas detected divided by the number of colonoscopies. Mean

adenoma per positive procedure (MAP+) will be defined as the total number of

adenoma detected divided by the number of colonoscopies in which at least one

adenoma is found. Mean additional adenomas detected beyond the first adenoma

per positive procedure (ADR-Plus) will be defined as the mean number of adenomas

detected after the first adenoma in procedures in which at least one adenoma is

found.

Lesions detected on the tandem right colon examination will be used for the

calculation of adenoma or polyp miss rate. Right colon AMR and hyperplastic polyp

miss rate (HPMR) will be calculated as the number of adenomas and hyperplastic

polyps missed in the first right colon examination divided by the total number of

adenoma and hyperplastic polyps detected during both the first and tandem right

colon examinations.

**Study Outcomes** 

The primary outcome is the right colon combined AMR and HPMR. Secondary

outcomes include right colon AMR, right colon HPMR, overall ADR, right colon ADR

and HPDR after the first examination, combined right colon ADR and HPDR after the

first and tandem examinations, overall advanced ADR, right colon advanced ADR,

overall MAP, right colon MAP, overall MAP+, right colon MAP+, overall ADR-Plus, and

right colon ADR-Plus. Procedure related parameters, including bowel cleansing,

insertion and withdrawal times, duration of tandem right colon examination, volume

of water infused and aspirated during insertion and withdrawal, and number of

abdominal compressions and/or position change, are also evaluated.

頁 8/13

## Sample size estimation

The sample size estimation is based on the assumption that WE colonoscopy reduces right colon combined AMR and HPMR compared to conventional CO2 insufflation colonoscopy. We estimate the overall right colon combined AMR and HPMR in the CO2 group to be 30% [30,31]. According to our previous study, the average detected number of right colon adenoma and hyperplastic polyp is <u>0.8 per subject after first right colon examination [32]</u>. To show a clinically important improvement of AMR reduction by the WE colonoscopy, we assume that WE colonoscopy should reduce the AMR by 15%. With a statistical power of 80% and a two-side significance level of 0.05, <u>131</u> patients will be needed in each study arm. To account for dropouts, incomplete procedures, and inadequate preparation, an additional 10% will be enrolled. Therefore, a total of <u>292</u> patients (<u>146</u> patients in each group) will be enrolled.

## Statistical analysis

Summary statistics will be presented as frequencies and percentages in the case of categorical variables and as the means with standard deviations (SD) in the case of continuous variables. Analysis will be performed by using an Intention-to-treat (ITT) approach. Interim analysis will be performed after enrollment of  $\underline{131}$  patients. Student's t-test for continuous factors, Wilcoxon rank sum test for ordinal variables (such as polyp size), and Chi-square test for categorical variables will be used to assess differences in demographic and clinical characteristics of patients in each group. Factors associated with adenoma detection by the first examiner will be identified by univariate analysis. Factors with a P value <0.1 on univariate analysis will be further entered into forward stepwise logistic regression analysis. The adjusted odds ratio with 95% confidence interval (CI) will be used to describe the

Date: 07/19/2019

influence of various factors on adenoma detection. All statistical analyses will be performed by using SAS version 9.3 or later (SAS Institute Inc., Cary, NC, USA). The criterion for statistical significance will be P value < 0.05.

## **REFERENCES:**

- 1. Dekker E, Rex DK. Advances in CRC prevention: screening and surveillance. Gastroenterology 2018;154:1970-1984.
- 2. Winawer SJ, Zauber AG, Nah M, et al. Prevention of colorectal cancer by colonoscopic polypectomy. N Engl J Med 1993;329:1977-1981.
- 3. Baxter NN, Warren JL, Barrett MJ, Stukel TA, Doria-Rose VP. Association between colonoscopy and colorectal cancer mortality in a US cohort according to site of cancer and colonoscopist specialty. J Clin Oncol 2012;30:2664-2669.
- 4. Nishihara R, Wu K, Lochhead P, et al. Long-term colorectal-cancer incidence and mortality after lower endoscopy. N Engl J Med 2013;369:1095-1105.
- 5. Doubeni CA, Weinmann S, Adams K, et al. Screening colonoscopy and risk for incident late-stage colorectal cancer diagnosis in average-risk adults: a nested case-control study. Ann Intern Med 2013;158:312-320.
- 6. le Clercq CM, Bouwens MW, Ronagh EJ, et al. Postcolonoscopy colorectal cancers are preventable: a population-based study. Gut 2014;63:957-963.
- 7. van Rijn JC, Reitsma JB, Stoker J, Bossuyt PM, van Deventer SJ, Dekker E. Polyp miss rate determined by tandem colonoscopy: a systemic review. Am J Gastroenterol 2006;101:343-350.
- 8. Leung FW, Harker JO, Jackson G, Okamoto KE, Behbahani OM, Jamgotchian NJ, Aharonian HS, Guth PH, Mann SK, Leung JW. A proof-of-principle prospective randomized controlled trial demonstrating improved outcomes in scheduled unsedated colonoscopy by the water method. Gastrointest Endosc

2010;72:693-700.

- Cadoni S, Gallittu P, Sanna S, Fanari V, Porcedda ML, Erriu M, Leung FW. A
  two-center randomized controlled trial of water-aided colonoscopy versus air
  insufflation colonoscopy. Endoscopy 2014;46:212-218.
- 10. Hsieh YH, Koo M, Leung FW. A patient-blinded randomized controlled trial comparing air insufflation, water immersion, and water exchange during minimally sedated colonoscopy. Am J Gastroenterol 2014;109:1390-1400.
- 11. Jia H, Pan Y, Guo X, et al. Water exchange method significantly improves adenoma detection rate: a multicenter randomized controlled trial. Am J Gastroenterol 2017;112:568-576.
- 12. Cadoni S, Falt P, Rondonotti E, et al. Water exchange for screening colonoscopy increases adenoma detection rate: a multicenter double-blinded randomized controlled trial. Endoscopy 2017;49:456-467.
- 13. Hsieh YH, Tseng CW, Hu CT, Koo M, Leung FW. Prospective multicenter randomized controlled trial comparing adenoma detection rate in colonoscopy using water exchange, water immersion, and air insufflation. Gastrointest Endosc 2017;86:192-201.
- 14. Fuccio L, Frazzoni L, Hassan C, La Marca M, Paci V, Smania V. et al. Water exchange colonoscopy increases adenoma detection rate: a systematic review with network meta-analysis of randomized controlled studies. Gastrointest Endosc 2018;88:589-597.
- 15. Jia H, Koo M, Hsieh YH, et al. Factors associated with adenoma detection in propofol-sedated patients. J Clin Gastroenterol 2019 (in press).
- 16. Leung FW, Koo M, Cadoni S, Falt P, Hsieh YH, Amato A, et al. Water exchange produces significantly higher adenoma detection rate than water immersion:

- pooled data from 2 multisite randomized controlled trials. J Clin Gastroenterol 2019 (in press).
- 17. Hsieh YH, Koo M, Tseng CW, et al. Reduction of multitasking distractions underlies the higher adenoma detection rate of water exchange compared to air insufflation blinded analysis of withdrawal phase videos. United European Gastroenterol J 2019 (in press).
- 18. Rondagh EJ, Bouwens MW, Riedl RG, et al. Endoscopic appearance of proximal colorectal neoplasms and potential implications for colonoscopy in cancer prevention. Gastrointest Endosc 2012;75:1218-1225.
- 19. Gupta S, Balasubramanian BA, Fu T, Genta RM, Rockey DC, Lash R. Polyps with advanced neoplasia are smaller in the right than in the left colon: implications for colorectal cancer screening. Clin Gastroenterol Hepatol 2012;10:1395-1401.
- 20. Leggett B, Whitehall V. Role of the serrated pathway in colorectal cancer pathogenesis. Gastroenterology 2010;138:2088-2100.
- 21. Rex DK, Ahnen DJ, Baron JA et al. Serrated lesions of the colorectum: review and recommendations from an expert panel. Am J Gastroenterol 2012;107:1315-1330.
- 22. Schreiner MA, Weiss DG, Lieberman DA. Proximal and large hyperplastic and nondysplastic serrated polyps detected by colonoscopy are associated with neoplasia. Gastroenterology 2010;139:1497-1502.
- 23. Hamoudah T, Ma K, Esteban M, et al. Patients with small and diminutive proximal hyperplastic polyps have higher rates of synchronous advanced neoplasia compared with patients without serrated lesions. Gastrointest Endosc 2018;87:1518-1526.
- 24. Jass JR. Hyperplastic polyps and colorectal cancer: Is there a link? Clin

- Gastroenterol Hepatol 2004;2:1-8.
- 25. Goldstein NS, Bhanot P, Odish E, Hunter S. Hyperplastic-like colon polyps that preceded microsatellite-unstable adenocarcinoma. Am J Clin Pathol 2003;119:778-796.
- 26. Lindholm CR, Anderson JC, Srivastava A. The dark side of the colon: current issues surrounding the significance, prevalence, detection, diagnosis and management of serrated polyps. Curr Opin Gastroenterol 2019;35:34-41.
- 27. Hetzel JT, Huang CS, Coukos JA, et al. Variation in the detection of serrated polyps in an average risk colorectal cancer screening cohort. Am J Gastroenterol 2010;105:2656-2664.
- 28. Wolf AMD, Fontham ETH, Church TR, et al. Colorectal cancer screening for average-risk adults: 2018 guideline update from the American Cancer Society. CA Cancer J Clin 2018;68:250-281.
- 29. Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc 2009;69:620-625.
- 30. Rex DK, Cutler CS, Lemmel GT, Rahmani EY, Clark DW, Helper DJ, et al. Colonoscopic miss rates of adenomas determined by back-to-back colonoscopies.

  Gastroenterology 1997;112:24-28.
- 31. Harrison M, Singh N, Rex DK. Impact of proximal colon retroflexion on adenoma miss rates. Am J Gastroenterol 2004;99:519-522.
- 32. Cheng CL, Kuo YL, Liu NJ. Tang JH, Fan JW, Lin CH, Tsui YN, Lee BP, Hung HL.

  Comparison of polyp detection during insertion and withdrawal versus only

  withdrawal of colonoscopy: a prospective randomized trial. J Gastroenterol

  Hepaptol 2019 (in press)